CLINICAL TRIAL: NCT02623829
Title: Botulinum Toxin is a Potential Prophylactic Therapy for Minimizing Post-excisional Scarring: A Double Blinded, Randomized Controlled Trial
Brief Title: Botulinum Toxin is a Potential Prophylactic Therapy for Minimizing Post-excisional Scarring (Allergan Botox Scar Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Daniel Michael Bernstein, Daniel Bernstein, MD, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GCO 15-1093
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Post-operative Excessive Scarring
Keywords: scar prophylaxis; Botulinum Toxin
MeSH Terms: interventions — Botulinum Toxins; Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin (Experimental): 50 units of botulinum toxin diluted in 1ml of normal saline will be administered. The forehead will be injected with 12, evenly spaced and symmetrical aliquots of 0.05ml(2.5 units) and the glabella will be injected at the nasal root and the medial aspect of the corrugators with 0.1ml(5 units) each in addition to the lateral aspect of each corrugator with 0.05ml(2.5 units). The injections will be administered with a 30G needle perpendicular to the skin.
  Interventions: Drug: Botulinum Toxin
- Saline (Sham Comparator): 1ml of normal saline will be injected with 12, evenly spaced and symmetrical aliquots of 0.05ml and the glabella will be injected at the nasal root and the medial aspect of the corrugators with 0.1ml each in addition to the lateral aspect of each corrugator with 0.05ml. The injections will be administered with a 30G needle perpendicular to the skin.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin — 50 units of botulinum toxin diluted in 1ml of normal saline will be administered.
  Other Names: Botox,; OnabotulinumtoxinA
  Arms: Botulinum Toxin
Drug: Saline — 1ml of normal saline will be administered
  Other Names: placebo
  Arms: Saline

SUMMARY:
Dermatological surgeons wear many hats to care for subjects with skin cancer. While their role in cancerous tissue removal results in superior cure rates, there is also a need for skilled excisional repair and effective wound healing regimens so the subject can heal with the least amount of scarring necessary. As such, numerous techniques have been developed for reducing the morbidity associated with excessive scarring. Various flaps and grafts allow the surgeon to approximate skin texture, thickness and adnexa with respect to the residual surrounding tissue. Optimal cosmetic and functional outcomes require close wound approximation with minimal static tension along the wound edge. In addition, there are post-operative wound care techniques that range from special dressings to cosmetic scar modification. To date, most surgical wounds are allowed to heal at least partially before scar revision or modulation is attempted.

Botulinum toxin presents a unique opportunity for surgeons to affect scar formation throughout the duration of the healing process. These effects are likely independent and adjunctive to any and all wound care techniques, and are primarily attributed to a reduction in dynamic tension on the wound edges. Most importantly, botulinum toxin's one time dosing requirements with respect to reduced scar formation precludes the variance inherent to standard wound care practices.

Therefore, it has been proposed that for selected subjects, botulinum toxin may be a safe, effective and reliable means for improved post-excisional repair outcomes. Botulinum toxin has been investigated as an inhibitor of excessive, post-excisional scar formation in plastic surgery and Otorhinolaryngology literature. However, these promising studies have yet to combine objective assessment measures of human scar formation in a randomized controlled trial. In addition, there are currently no formal studies of botulinum toxin as a prophylactic against excess scarring in the dermatological literature. Fortunately, Botulinum toxin dosing in the forehead for the purposes of inhibiting excessive scar formation is comparable to the amount given for cosmetic purposes, which is commonplace in dermatology and well-studied.

DETAILED DESCRIPTION:
This study will attempt to assess the efficacy of Botulinum toxin as a prophylactic treatment in post-excisional repairs for the purpose of preventing excess scar formation. The end points will be the evaluation of each scar using the Manchester Scar Scale.

All MSS and mMSS assessments will be performed in a standardized fashion. The mMSS assessments will be blinded and performed by board-certified dermatologists in the Department of Dermatology, Faculty Practice Associates, Icahn School of Medicine at Mount Sinai, New York City.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults at least 18 years old.
* Subjects must be scheduled for an excision of forehead skin due to any etiology, with a same day, single stage closure planned as the most likely surgical repair.
* Subjects must be able to read, sign, and understand the informed consent.
* Subject is willing and able to participate in the study as an outpatient, making several visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subjects with an unstable medical condition as deemed by the clinical investigator, including review of the subject's prior and current medications.
* Subjects with Myasthenia gravis, Lambert-Eaton Syndrome or other neuromuscular disorder.
* Subjects taking medications that may alter the function of neuromuscular junctions (i.e. aminoglycoside antibiotics)
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have a history of keloids.
* Known allergy to botulinum toxin.
* Subjects who are not able to be closed with a same day, single stage technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Michael Bernstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinia, New York, New York, United States

REFERENCES:
- [Background] Jablonka EM, Sherris DA, Gassner HG. Botulinum toxin to minimize facial scarring. Facial Plast Surg. 2012 Oct;28(5):525-35. doi: 10.1055/s-0032-1325641. Epub 2012 Oct 1. PMID 23027220
- [Background] Gassner HG, Brissett AE, Otley CC, Boahene DK, Boggust AJ, Weaver AL, Sherris DA. Botulinum toxin to improve facial wound healing: A prospective, blinded, placebo-controlled study. Mayo Clin Proc. 2006 Aug;81(8):1023-8. doi: 10.4065/81.8.1023. PMID 16901024
- [Background] Gassner HG, Sherris DA, Otley CC. Treatment of facial wounds with botulinum toxin A improves cosmetic outcome in primates. Plast Reconstr Surg. 2000 May;105(6):1948-53; discussion 1954-5. doi: 10.1097/00006534-200005000-00005. PMID 10839391
- [Background] Sherris DA, Gassner HG. Botulinum toxin to minimize facial scarring. Facial Plast Surg. 2002 Feb;18(1):35-9. doi: 10.1055/s-2002-19825. PMID 11823931
- [Background] Gassner HG, Sherris DA, Friedman O. Botulinum toxin-induced immobilization of lower facial wounds. Arch Facial Plast Surg. 2009 Mar-Apr;11(2):140-2. doi: 10.1001/archfacial.2009.3. No abstract available. PMID 19289689
- [Background] Carruthers J, Fagien S, Matarasso SL; Botox Consensus Group. Consensus recommendations on the use of botulinum toxin type a in facial aesthetics. Plast Reconstr Surg. 2004 Nov;114(6 Suppl):1S-22S. doi: 10.1097/01.PRS.0000144795.76040.D3. PMID 15507786
- [Background] Carruthers A, Carruthers J, Cohen J. A prospective, double-blind, randomized, parallel- group, dose-ranging study of botulinum toxin type a in female subjects with horizontal forehead rhytides. Dermatol Surg. 2003 May;29(5):461-7. doi: 10.1046/j.1524-4725.2003.29114.x. PMID 12752512
- [Background] Zimbler MS, Nassif PS. Adjunctive applications for botulinum toxin in facial aesthetic surgery. Facial Plast Surg Clin North Am. 2003 Nov;11(4):477-82. doi: 10.1016/S1064-7406(03)00071-3. PMID 15062252
- [Background] Beausang E, Floyd H, Dunn KW, Orton CI, Ferguson MW. A new quantitative scale for clinical scar assessment. Plast Reconstr Surg. 1998 Nov;102(6):1954-61. doi: 10.1097/00006534-199811000-00022. PMID 9810991
- [Background] Duncan JAL, Bond JS, Mason T, Ludlow A, Cridland P, O'Kane S, Ferguson MWJ. Visual analogue scale scoring and ranking: a suitable and sensitive method for assessing scar quality? Plast Reconstr Surg. 2006 Sep 15;118(4):909-918. doi: 10.1097/01.prs.0000232378.88776.b0. PMID 16980850
- [Background] Durani P, McGrouther DA, Ferguson MW. Current scales for assessing human scarring: a review. J Plast Reconstr Aesthet Surg. 2009 Jun;62(6):713-20. doi: 10.1016/j.bjps.2009.01.080. Epub 2009 Mar 20. PMID 19303834

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin: subcutaneous injections of onabotulinumtoxinA (1 mL = 50 units) immediately following closure of forehead wounds
- Saline: subcutaneous injections of saline (1 mL) immediately following closure of forehead wounds
Period: Overall Study
Arm/Group | Botulinum Toxin | Saline
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Saline | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [45 to 72] | 59 [43 to 75] | 58 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 20 | 40
Smoking history [Count of Participants; unit: Participants] | 2 | 2 | 4
Autoimmune conditions [Count of Participants; unit: Participants] | 1 | 1 | 2
Scar location [Count of Participants; unit: Participants]
  Median forehead | 2 | 2 | 4
  Paramedian forehead | 10 | 10 | 20
  Lateral forehead | 8 | 8 | 16
Scar length [Median (Inter-Quartile Range); unit: mm] | 58 [32 to 75] | 54 [28 to 72] | 55 [32 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Modified Manchester Scar Scale (MMSS) Score
Description: MMSS scores range 5-18, higher score indicates poorer health outcomes. The MMSS assesses color, texture, distortion and contour of the scar.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 8 [6 to 11] | 11.5 [9 to 14]

2. Secondary Outcome: Visual Analog Scar Scale
Description: Visual Analog Scar Scale (VASS), full score range 0-10 higher score indicates poorer health outcomes
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 2 [1 to 3] | 3.5 [2 to 4]

3. Secondary Outcome: Scar Width
Description: Scar width at 6 months after treatment
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 20 | 20
mm | 2.2 [1.8 to 3.0] | 3.2 [2.8 to 3.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Botulinum Toxin | Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin (N=20) | Saline (N=20)
mild unilateral eyelid ptosis (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT02623829/Prot_SAP_000.pdf